CLINICAL TRIAL: NCT05677100
Title: DRAIN-HF: Diuretics Alone vs. Aortix Endovascular Device for Acute Heart Failure
Brief Title: Diuretics Alone vs. Aortix Endovascular Device for Acute Heart Failure
Acronym: DRAIN-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Procyrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP001
Record Dates: First submitted 2022-10-07; First posted 2023-01-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Cardiorenal Syndrome; Cardio-Renal Syndrome; ADHF; Heart Failure, Systolic; Heart Failure, Diastolic; Heart Failure; With Decompensation; Heart Failure, Congestive
Keywords: mechanical circulatory support; percutaneous
MeSH Terms: conditions — Heart Failure; Cardio-Renal Syndrome; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: The patients will be randomized 1:1 and will be receiving their treatment in parallel to each other. An additional non-randomized registry is also included
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Treatment Arm (Experimental): Eligible ADHF patients with diuretic resistance (irrespective of ejection fraction) will be enrolled and randomized 1:1 to either the Aortix system or standard of care medical management. Randomization will be stratified by ejection fraction.
  Interventions: Device: Aortix System
- Control Arm (No Intervention): The Control arm should receive standard of care therapy as per the study directed Diuretic Care Treatment Algorithm.
- Advanced HF Registry (Experimental): For the Advanced HF registry, all eligible enrolled subjects will receive Aortix system support.
  Interventions: Device: Aortix System

INTERVENTIONS:
Device: Aortix System — Aortix is a circulatory support device for chronic heart failure patients on medical management who have been hospitalized for acute decompensated heart failure (ADHF) and are resistant to diuretic therapy.
  Other Names: Aortix Pump
  Arms: Advanced HF Registry; Treatment Arm

SUMMARY:
Aortix is a circulatory support device for chronic heart failure patients on medical management who have been hospitalized for acute decompensated heart failure (ADHF) and have persistent congestion despite usual medical therapy.

Eligible ADHF patients with diuretic resistance (irrespective of ejection fraction) will be enrolled and randomized 1:1 to either the Aortix system or standard of care medical management.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, randomized, nonblinded study to evaluate the safety and effectiveness of the Aortix System versus standard of care medical therapy in patients hospitalized with acute decompensated heart failure (ADHF) and persistent congestion despite usual medical management.Eligible ADHF patients with diuretic resistance (irrespective of ejection fraction) will be enrolled and randomized 1:1 to either the Aortix system or standard of care medical management. Randomization will be stratified by ejection fraction..

An additional registry arm will enroll patients who are considered candidates for advanced therapies in the near-term, but need improvement in their renal function to be able to receive additional medical therapies. All eligible enrolled registry subjects will receive Aortix system support.

Planned study population is male or female patients 21 years of age or greater, with acute decompensated heart failure and diuretic resistance who remain congested despite standard of care medical therapy.

This study will enroll up to 295 subjects with heart failure at 45 clinical sites in the United States and up to 5 OUS sites. The randomized study includes up to 215 subjects and the Advanced HF registry includes up to 80 subjects.

ELIGIBILITY:
Inclusion Criteria (Randomized Study):

* Currently admitted to the hospital with a primary diagnosis of decompensated heart failure, irrespective of ejection fraction (EF);
* Patients should be on maximally tolerated diuretic therapy and not diuresing sufficiently before being enrolled in DRAIN-HF. After being up-titrated on diuretics, patients should be followed for at least 24 hours on the higher of: i) furosemide 80 mg IV bid or equivalent or ii) IV furosemide or equivalent IV loop diuretic at a dose 2.5 x total daily home dose of furosemide equivalents in 2 divided doses, as tolerated, patient must have: Urine Output <1,500mL in a 12-hour period OR a Net Fluid Loss ≤375mL in a 12-hour period.
* Persistent signs and/or symptoms of congestion as evidenced by at least 2+ pitting edema, elevated jugular venous pressure >12 cm water or ascites after treatment with IV diuretics per inclusion criterion 2.;
* Age >21 years and able to provide written informed consent;
* Negative pregnancy test if patient is of child-bearing potential.

Exclusion Criteria (Randomized Study):

* Treatment with high dose IV inotropes within the last 48 hours prior to enrollment. High dose is defined as >5 µg/kg/min dopamine OR >5 µg/kg/min dobutamine OR >0.375 µg/kg/min milrinone;
* Active and ongoing hypotension with a systolic blood pressure <90 mmHg lasting more than 30 minutes or a mean arterial pressure (MAP) <60 mmHg lasting more than 30 minutes at enrollment;
* Treatment with vasopressors (defined as phenylephrine, norepinephrine, epinephrine or, vasopressin) within 48 hours prior to enrollment;
* An estimated PASP of >80 mmHg as measured on echocardiogram or echocardiographic evidence of primarily right heart failure;
* Treatment with IV diuretics (does not have to be continuous) for ≥21 days during the current hospitalization (including time spent at an outside hospital);
* Acute kidney failure defined as an increase in serum creatinine to ≥4.0mg/dL (≥353.6 µmol/L) at enrollment;
* Evidence of contrast induced nephropathy, nephritis or nephrotic syndrome;
* Prior kidney transplant, single kidney, partial nephrectomy OR use of dialysis, continuous renal replacement therapy (CRRT) or ultrafiltration in the last 90 days prior to enrollment;
* Confirmed decompensated cirrhosis (defined as Child Pugh class B or C) or concern for shock liver (AST > 1000U/L or total Bilirubin > 5.0mg/dl) at enrollment;
* Presence of an active, uncontrolled infection that would preclude safe placement or removal of the device;
* Prior heart transplant or likely heart transplantation before the 30- day follow-up visit;
* Current or previous support with a durable LVAD at any time or planned LVAD insertion before the 30-day follow-up visit;
* Use of an intra-aortic balloon pump (IABP), extracorporeal membrane oxygenation (ECMO), or percutaneous ventricular assist devices (e.g. Impella or TandemHeart) within the last 30 days;
* Known amyloidosis of any type;
* Acute myocardial infarction Type 1 within 30 days of enrollment, or planned coronary revascularization in the next 30 days;
* Stroke within 30 days of enrollment;
* Severe Bleeding Risk (any of the following):

  1. Previous intracranial bleed unless there is documentation in the medical record (from a physician that is not part of the study) that the patient can safely use anticoagulation for 7 days,
  2. GI bleeding within 6 months requiring hospitalization and/or transfusion,
  3. Recent major surgery within 30 days if the surgical wound is judged to be associated with an increased risk of bleeding,
  4. Procedure with arterial ilio-femoral access > 6 FR within 30 days,
  5. Platelet count <75,000 cells/mm3,
  6. Uncorrectable bleeding diathesis or coagulopathy (e.g. INR ≥2 not due to anticoagulation therapy) or hypercoaguable state including HIT;
  7. Inability to tolerate anticoagulation therapy for up to 7 days.
* Contraindicated Anatomy :

  1. Descending aortic anatomy that would prevent safe placement of the device [<18 mm or >31 mm aorta diameter at deployment location (measured between the superior aspect of the T10 vertebra and superior aspect of the L1 vertebra)],
  2. Ilio-femoral diameter or peripheral vascular anatomy that would preclude safe placement of a 21F (outer diameter) introducer sheath,
  3. Femoral artery depth inconsistent with use of closure device,
  4. Abnormalities or severe vascular disease that would preclude safe access and device delivery (e.g. aneurysm with thrombus, marked tortuosity, significant narrowing or inadequate size of the abdominal aorta, iliac or femoral arteries, or severe calcification),
  5. Known connective tissue disorder (e.g. Marfan Syndrome) or other aortopathy at risk of vascular injury,
  6. Any endovascular stent graft in the descending aorta. Any endovascular stent graft in the femoro-iliac vessels that is not well endothelialized and would preclude safe introduction/removal of the Aortix pump as demonstrated by imaging.
* Known hypersensitivity or contraindication to study or procedure medications (e.g. anticoagulation therapy) or device materials (e.g. history of severe reaction to nickel or nitinol);
* Participation in any other clinical investigation that is likely to confound study results or affect the study;
* Poor health such that the patient is unable to undergo the Aortix device placement/retrieval and/or unlikely to be able to survive to the 30-day visit;
* Unable or unwilling to undergo screening (imaging, PA Catheter placement), device implant and retrieval procedures or return for 30-day visit.

Inclusion Criteria (Advanced Heart Failure Registry):

* Currently admitted to the hospital with a primary diagnosis of decompensated HF, irrespective of ejection fraction (EF).
* Patient has already been evaluated and indicated to receive an LVAD or heart transplant and will receive the LVAD or be listed for heart transplantation in the next 30 days if their congestion status and renal function improves.
* Patient must have been treated with ≥ 80 mg IV furosemide bid or equivalent and have evidence of increasing diuretic dosing requirements over the past 12 months, as tolerated.
* Must have evidence of refractoriness to medical management as documented by persistent signs and/or symptoms of congestion as evidenced by at least 2+ pitting edema, elevated jugular venous pressure >12 cm water, or ascites after treatment with IV diuretics for a minimum of 24 hours.
* Serum creatinine ≥ 2.0 mg/dL AND eGFR ≤ 45 ml/min/1.73m2 at time of enrollment
* Age ≥ 21 years and able to provide written informed consent.
* Negative pregnancy test if patient is of childbearing potential.

Exclusion Criteria (Advanced Heart Failure Registry):

* Treatment with high dose IV inotropes within 48 hours prior to enrollment. High dose is defined as any one of the following: >5 µg/kg/min dopamine OR >5 µg/kg/min dobutamine OR >0.375 µg/kg/min milrinone.
* Active and ongoing hypotension with a systolic blood pressure <80 mmHg lasting more than 30 minutes or a mean arterial pressure (MAP) <55 mmHg lasting more than 30 minutes at enrollment.
* Treatment with vasopressors (defined as phenylephrine, norepinephrine, epinephrine or, vasopressin) within 48 hours prior to enrollment.
* An estimated PASP of >80 mmHg as measured on echocardiogram or echocardiographic evidence of primarily right heart failure.
* Acute kidney failure defined as an increase in serum creatinine to ≥ 4.0mg/dL at enrollment.
* Evidence of contrast-induced nephropathy, nephritis, or nephrotic syndrome.
* Prior kidney transplant, single kidney, partial nephrectomy OR use of dialysis, continuous renal replacement therapy (CRRT), or ultrafiltration in the last 90 days prior to enrollment.
* Confirmed decompensated cirrhosis (defined as Child Pugh class B or C) or concern for shock liver (AST > 1000U/L or total Bilirubin > 5.0mg/dl) at enrollment.
* Presence of an active, uncontrolled infection that would preclude safe placement or removal of the device.
* Current or previous support with a durable LVAD.
* INTERMACS Profile 1 at enrollment.
* Currently on mechanical ventilatory support.
* Use of an intra-aortic balloon pump (IABP) within the last 14 days or use of an extracorporeal membrane oxygenation (ECMO) or percutaneous ventricular assist device (e.g., Impella or TandemHeart) within the last 30 days.
* Known amyloidosis of any type.
* Acute myocardial infarction Type 1 within 30 days of enrollment or planned coronary revascularization in the next 30 days.
* Stroke within 30 days of enrollment.
* Severe Bleeding Risk (any of the following):

  * Previous intracranial bleed unless there is documentation in the medical record (from a physician that is not part of the study) that the patient can safely use anticoagulation for 7 days.
  * GI bleeding within 6 months requiring hospitalization and/or transfusion.
  * Recent major surgery within 30 days if the surgical wound is judged to be associated with an increased risk of bleeding.
  * Procedure with arterial ilio-femoral access > 6 Fr within 30 days.
  * Platelet count <75,000 cells/mm3 .
  * Uncorrectable bleeding diathesis or coagulopathy (e.g., INR≥ 2 not due to anticoagulation therapy) or hypercoagulable state including HIT.
  * Inability to tolerate anticoagulation therapy for up to 7 days.
* Contraindicated Anatomy :

  * Descending aortic anatomy that would prevent safe placement of the device [<18 mm or >31 mm aorta diameter at deployment location (measured between the superior aspect of the T10 vertebra and superior aspect of the L1 vertebra)].
  * Ilio-femoral diameter or peripheral vascular anatomy that would preclude safe placement of a 21 Fr (outer diameter) introducer sheath.
  * Femoral artery depth inconsistent with use of closure device.
  * Abnormalities or severe vascular disease that would preclude safe access and device delivery (e.g., aneurysm with thrombus; marked tortuosity; significant narrowing or inadequate size of the abdominal aorta, iliac, or femoral arteries; or severe calcification).
  * Known connective tissue disorder (e.g., Marfan Syndrome) or other aortopathy at risk of vascular injury.
  * Any endovascular stent graft in the descending aorta. Any endovascular stent graft in the femoro-iliac vessels that is not well endothelialized and would preclude safe introduction/removal of the Aortix pump as demonstrated by imaging.
* Known hypersensitivity or contraindication to study or procedure medications (e.g., anticoagulation therapy) or device materials (e.g., history of severe reaction to nickel or nitinol).
* Participation in any other clinical investigation that is likely to confound study results or affect the study.
* Poor health such that the patient is unable to undergo the Aortix device placement/retrieval and/or unlikely to be able to survive to the 30-day visit.
* Unable or unwilling to undergo screening, device implant and retrieval procedures, or return for 30-day visit.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Incidence of Aortix Device / Procedural-Related Major Adverse Events (MAE) through 30 days of Follow-up. | Baseline to 30 day Follow-Up
  Incidence of Major Adverse Events
Primary Effectiveness Endpoint: Combined composite of clinically significant reduction in net fluid loss over 7 days and freedom from mortality or heart failure re-hospitalization/therapy escalation from the baseline visit to the 30-day follow-up visit. | Baseline to 30 day Follow-Up
  Composite of net fluid loss, mortality and HF hospitalization/escalation of therapy

SECONDARY OUTCOMES:
Net Fluid Loss | Baseline to Day 7
  Change in Net Fluid Loss from Baseline to Day 7/Discharge
All-cause Mortality | Baseline to 30 day Follow-Up
  Rate of mortality
HF Re-Hospitalization or escalation of HF therapy | Baseline to 30 day Follow-Up
  Evaluation of HF re-hospitalization and therapy escalation
eGFR | Baseline to 30 day Follow-Up
  Evaluation of changes in eGFR
NT-proBNP | Baseline to 30 day Follow-Up
  Evaluation of NT-proBNP
Patient Reported Dyspnea Assessment | Baseline to 30 day Follow-Up
  Change in patient reported dyspnea scale
Standing body weight | Baseline to 30 day Follow-Up
  Change in standing body weight
Incidence and percentages of major adverse events (MAE) Pooled | Baseline to 30 day Follow-Up
  Incidence and percentages of major adverse events (MAE) pooled analysis of Aortix randomized cohort and registry cohort

CONTACTS AND LOCATIONS:
Locations (47):
- United States (46):
  - Banner--University Medical Center Phoenix, Phoenix, Arizona
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - HonorHealth Medical Center, Scottsdale, Arizona
  - John Muir Health, Concord, California
  - Zuckerberg San Francisco General, San Francisco, California
  - San Francisco Veterans Administration, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Ascension Sacred Heart, Pensacola, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - BayCare Medical/St. Joseph's Hospital, Tampa, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Healthcare Inc., Augusta, Georgia
  - Wellstar Research Institue, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate IMMC, Chicago, Illinois
  - Advocate Aurora - Good Samaritan, Downers Grove, Illinois
  - Ascension via Christi Kansas, Wichita, Kansas
  - University of Michigan, Cardiovascular Medicine, Ann Arbor, Michigan
  - Henry Ford, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Presbyterian - Brooklyn Methodist Hospital, Brooklyn, New York
  - Mount Sinai Morningside, New York, New York
  - Nyph/Cumc, New York, New York
  - Northwell Health (Lenox Hill), New York, New York
  - Nuvance Health, Poughkeepsie, New York
  - Northwell Health (Staten Island), Staten Island, New York
  - Atrium Health Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Fort Worth, Texas
  - Texas Heart Institute, Houston, Texas
  - Baylor Scott & White, Plano, Texas
  - Intermountain Health, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No